CLINICAL TRIAL: NCT00052832
Title: Phase II Study of Doxercalciferol for the Treatment of Myelodysplastic Syndromes
Brief Title: Doxercalciferol in Treating Patients With Myelodysplastic Syndrome or Chronic Myelomonocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: HO02403; P30CA014520 (NIH); HO02403 (Other: University of Wisconsin Carbone Cancer Center); 2002-184 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH/MEDICINE (Other: UW Madison)
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2015-09

CONDITIONS: Leukemia; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: chronic myelomonocytic leukemia; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; de novo myelodysplastic syndromes; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders | interventions — 1 alpha-hydroxyergocalciferol

INTERVENTIONS:
Dietary Supplement: doxercalciferol

SUMMARY:
RATIONALE: Doxercalciferol may improve low blood cell counts and decrease the need for blood transfusions and may be an effective treatment for myelodysplastic syndrome or chronic myelomonocytic leukemia.

PURPOSE: Phase II trial to study the effectiveness of doxercalciferol in treating patients who have myelodysplastic syndrome or chronic myelomonocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate of patients with myelodysplastic syndromes or chronic myelomonocytic leukemia treated with doxercalciferol.
* Determine the toxicity profile of this drug in these patients.
* Determine the time to progression and overall survival of patients treated with this drug.

OUTLINE: Patients receive oral doxercalciferol daily for 12 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: Approximately 41 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Morphologically and cytogenetically confirmed myelodysplastic syndromes or chronic myelomonocytic leukemia

  * No more than 20% blasts by bone marrow biopsy
* Must meet at least 1 of the following criteria:

  * Anemia

    * Hemoglobin less than 11 g/dL over a 2-month period
  * Thrombocytopenia
  * Neutropenia

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics

Hepatic

* ALT and AST less than 1.5 times upper limit of normal
* Bilirubin less than 3 mg/dL
* Albumin greater than 3.0 g/dL

Renal

* Creatinine clearance greater than 50 mL/min
* No history of hypercalcemia
* No renal stones within the past 5 years

Cardiovascular

* No clinically significant heart failure
* No uncontrolled hypertension

Pulmonary

* No clinically significant pulmonary failure

Other

* Not pregnant
* Fertile patients must use effective contraception during and for 6 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 4 weeks since prior growth factor or cytokine therapy

Chemotherapy

* At least 8 weeks since prior cytotoxic chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* Concurrent transfusion support allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-09; Primary Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark B. Juckett, MD, Study Chair — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- [Result] Petrich A, Kahl B, Bailey H, Kim K, Turman N, Juckett M. Phase II study of doxercalciferol for the treatment of myelodysplastic syndrome. Leuk Lymphoma. 2008 Jan;49(1):57-61. doi: 10.1080/10428190701713648. PMID 18203012
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu